CLINICAL TRIAL: NCT06299345
Title: The Effect of Motor Imagery Dosage on Motor Learning in Healthy Adults, A Pilot Study
Brief Title: The Effect of Motor Imagery Dosage on Motor Learning in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmed Mahmoud Kadry (Other)
Collaborators: Concordia University Wisconsin (Other)
Responsible Party: Sponsor-Investigator, Ahmed Mahmoud Kadry, Associate Professor of Physical Therapy, Kafrelsheikh University
Organization: Kafrelsheikh University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1870394-1
Record Dates: First submitted 2024-02-18; First posted 2024-03-07 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Healthy
Keywords: Motor Imagery; Dosage; Motor Learning

STUDY DESIGN:
Who Masked: Participant
Masking Description: The participants were blinded about which group they were allocated (control or intervention)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (CG) (Sham Comparator): Physically performed the task once per session. No MI. The physical task is a mirror tracing game that requires participants to trace a star shape viewed through a mirror, going as fast as possible while staying within the lines.
  Interventions: Other: NO motor imagery training
- low-dose group (LD) (Experimental): In addition to physically performing the motor task once in session 1, then they performed MI for 6 minutes (2 min x 3 sets) per session. MI for this study took the form of non-guided first-person mental practice. First-person imagery was explained to each participant where they imagined performing the target skill through their own eyes rather than if they were a bystander watching someone else do the task (third person).
  Interventions: Other: Motor imagery training
- high-dose group (HD) (Experimental): In addition to physically performing the motor task once in session 1, then MI for 12 minutes (2 min x 6 sets) per session. The MI technique was the same as the LD group.
  Interventions: Other: Motor imagery training

INTERVENTIONS:
Other: Motor imagery training — MI for this study took the form of non-guided first-person mental practice. First-person imagery was explained to each participant where they imagined performing the target skill through their own eyes rather than if they were a bystander watching someone else do the task (third person).
  Arms: high-dose group (HD); low-dose group (LD)
Other: NO motor imagery training — The participants performed the physical task only. It is a mirror tracing game that requires participants to trace a star shape viewed through a mirror, going as fast as possible while staying within the lines.
  Arms: control group (CG)

SUMMARY:
The goal of this clinical trial is to compare the effects of different durations of Motor Imagery (MI) practice and physical practice on motor performance enhancement in healthy adults. The main questions it aims to answer are:

* Does Motor Imagery (MI) practice improve motor performance?
* How do different doses of MI practice (low vs. high) compare to no MI practice in enhancing motor performance?

Participants:

* Be randomly assigned to one of three groups: no MI practice (control group), low dose MI practice (6 minutes per session), or high dose MI practice (12 minutes per session).
* Complete nine sessions over three weeks, practicing a timed mirror tracing task.
* Have their performance measured in each session by the time taken to complete the task and the number of errors made.

Compared the control group, low dose MI group, and high dose MI group to see if there are significant differences in motor performance enhancement, aiming to determine the effectiveness of MI and the optimal dose for practice.

ELIGIBILITY:
Inclusion Criteria:

* no history of motor dysfunction, coordination disorders, or surgical procedures in the past 6 months
* scored 4 or less on the Movement Imagery Questionnaire (MIQ) on the non-dominant hand.

Exclusion Criteria:

* Played the target task in the past 6 months
* Subjects were ambidextrous

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-04-28 (Actual)

PRIMARY OUTCOMES:
Time | Time was measured at the end of each session, with intervals of 3 session/week for 3 weeks with total of 9 sessions. So, the research ended up with 9 reading for the time.
  The time to complete the physical tracing task was measured from when the investigator said 'GO' until the participant returned the pen to the starting point. The physical tracing task is a mirror tracing game that requires participants to trace a star shape viewed through a mirror, going as fast as possible while staying within the lines.
Errors | Errors were counted at the end of each session, with intervals of 3 session/week for 3 weeks with total of 9 sessions. So, the research ended up with 9 reading for the time.
  Errors were operationally defined as each time the pen went outside of the shape lines while doing the physical tracing task. Crossing a line and returning to the original trace was counted as one error. Errors were counted by the number of times the pen went outside the lines.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Kadry, PhD, Principal Investigator — Associate Professor of Physical Therapy, Kafrelsheikh University
Locations (2):
- Concordia University Wisconsin, Mequon, Wisconsin, United States
- Kafrelshaikh University, Kafr ash Shaykh, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data from this study, including individual participant data (IPD) and associated documentation, will be made available upon reasonable request to the principal investigator. Requests will be considered when accompanied by a detailed proposal, including a clear justification for the use of the data. Such requests will be subject to a review process to ensure compatibility with participant consent and the ethical guidelines governing the study. Data sharing will be facilitated under a data use agreement that specifies the terms and conditions to ensure the privacy and confidentiality of participants
Supporting Information: Study Protocol, SAP
Time Frame: 1 year from publication
Access Criteria: upon request from the principal investigator with appropriate justification